CLINICAL TRIAL: NCT03578575
Title: To Investigate the Molecular Mechanism of Traditional Chinese Medicine Constitution Using Next-generation Sequencing in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH106-REC1-068
Record Dates: First submitted 2018-05-16; First posted 2018-07-06 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Concurrent chemo-radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — danggui buxue decoction

STUDY DESIGN:
Intervention Model Description: 120 subjects are divided into experimental group and control group (placebo).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danggui Buxue Tang group (Experimental): Use Danggui Buxue Tang 5g/time, 3 times a day, for 12 weeks.
  Interventions: Drug: Danggui Buxue Tang
- Placebo group (Placebo Comparator): Use Placebo 5g/time, 3 times a day, for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danggui Buxue Tang — Danggui Buxue Tang is an extracted powder of traditional Chinese medicine formula.
  Arms: Danggui Buxue Tang group
Drug: Placebo — Placebo is a very low dose Danggui Buxue Tang powder.
  Arms: Placebo group

SUMMARY:
To investigate the molecular mechanism of traditional Chinese medicine constitution, the investigators proposed a randomized, double-blind, placebo-controlled, phase II trial to recruit 120 patients with nasopharyngeal cancer. Next generation sequencing, immune repertoire, gut microbiota, traditional Chinese medicine constitution and tongue diagnosis would be examined before/after 16 weeks of treatment of Danggui Buxue Tang from the beginning of concurrent chemoradiotherapy in this project. The correlation between different examinations would be analyzed to investigate the molecular mechanism of traditional Chinese medicine constitution. Disease survival, recurrence, and quality of life would be also followed up for two years to evaluate the benefit of Danggui BuxueTang.

DETAILED DESCRIPTION:
The basis for academic excellence is the interdisciplinary cooperation. The individualized medicine is the future trends, and the theory of body constitution is the most potential study for the individualized medicine and to research the process and prognosis of disease. Technique of next-generation sequencing (NGS) is also involved to comprehend to the mechanism of the prescriptions under the theory of body constitution.

The nasopharyngeal cancer is a Chinese-specific disease, and radiation therapy has remarkable effect. There are many studies proving that Traditional Chinese medication can relieve the side effect of radiation therapy. The study will combine next-generation sequencing and TCM diagnostic tool, and analyze the transformation of body constitution and the performance of genes related to radiation therapy. The results may reveal the molecular mechanism of TCM constitutions and the benefit of Danggui BuxueTang, and may be used for early screen and prevention to other cancers or diseases. Furthermore, it can help to develop the potential drugs.

The study plans to collect 120 cases within two years. The participants would be divided randomly to the experimental group and control group. The blood sample would be taken for next generation sequencing analysis before the radiation therapy, and after the radiation therapy combined with traditional Chinese medication. The result of samples would be compared with each other to identify "Qi deficiency gene" and "TCM effective gene".

ELIGIBILITY:
Inclusion Criteria:

Patients with pathological diagnosis of nasopharyngeal carcinoma stage II ~ IVa (AJCC eighth edition) preparing to receive concurrent chemoradiotherapy

Exclusion Criteria:

* Pregnant or lactating women
* ECOG PS (ECOG performance status) scores of over 2 points for each day's performance assessment
* Take anticoagulants or antiplatelet agents such as aspirin, warfarin, etc.
* Cannot accept routine treatment, or can not cooperate with the research program

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between next-generation sequencing analysis and traditional Chinese medicine constitution | The biomarker as assessed by Next-generation sequencing analysis, Change from baseline in the gene expression at 16 weeks of treatment of Danggui Buxue Tang from the beginning of concurrent chemoradiotherapy and 2-year follow-up.
  Identification of biomarkers by next-generation sequencing analysis in nasopharyngeal cancer patients.

SECONDARY OUTCOMES:
The quality of life as assessed by the score of questionnaire of European Organisation for Research and Treatment of Cancer C30 | Change from baseline in score of questionnaire at 16 weeks of treatment of Danggui Buxue Tang from the beginning of concurrent chemoradiotherapy and 2-year follow-up.
  The quality of life for cancer patients as assessed by the score of cancer-specific questionnaire, "European Organisation for Research and Treatment of Cancer (EORTC C30)", which is cancer-specific core questionnaire for use in various cancers with 30 in Functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures etc), with range from 1 (Not at all) to 4 (Very much), and from 1 (Very poor) to 7 (Excellent), scoring from 0 to 100. For functional and global quality of life scales, higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
The quality of life as assessed by the score of questionnaire of European Organisation for Research and Treatment of Cancer H&N35 | Change from baseline in score of questionnaire at 16 weeks of treatment of Danggui Buxue Tang from the beginning of concurrent chemoradiotherapy and 2-year follow-up.
  The quality of life as assessed by the score of a head & neck cancer-specific questionnaire, "European Organisation for Research and Treatment of Cancer Head and Neck Module (EORTC H&N35)", with 35 items to evaluate symptoms encountered by patients with head and neck cancer in 18 domains, including in 7 multiple-item scales (Pain, Swallowing, Senses, Speech, Social eating, Social contact, and Sexuality) and 11 single items (eg, Opening mouth, Sticky saliva, Dry mouth, etc), with range from 1 (Not at all) to 4 (Very much), and from 1 (Very poor) to 7 (Excellent). EORTC H&N35)have standardized scores ranging from 0 to 100, with higher scores indicating a greater degree of symptoms.
Survival rate | throughout the study, an average of 2 year
  Survival after treatment
Disease recurrence | throughout the study, an average of 2 year
  Disease recurrence after treatment
Next-generation sequencing | pre-treatment and after 16 weeks of treatment
  The comparison of next-generation sequencing of human gene analysis after treatment
Immune repertoire | pre-treatment and after 16 weeks of treatment
  The comparison of IgG, IgA and T cell receptor immune repertoire after treatment
Microbiota | pre-treatment and after 16 weeks of treatment
  The comparison of gut microbiota after treatment
Tongue diagnosis | pre-treatment and after 16 weeks of treatment
  The comparison of Tongue diagnosis after treatment
Constitution in Chinese Medicine Questionnaire (CCMQ) | Change from baseline in score of questionnaire at 16 weeks of treatment of Danggui Buxue Tang from the beginning of concurrent chemoradiotherapy and 2-year follow-up.
  The Chinese medicine constitution as assessed by the score of Constitution in Chinese Medicine Questionnaire, consists of 60 items in 9 types of Chinese medicine constitution, gentleness, Qi-deficiency, Yang-deficiency, Yin-deficiency, phlegm-dampness, dampness-heat, blood-stasis, Qi-stagnation, and special diathesis, with scaling range from 1(None) to 5(Always). The score would be transform to adjusted scores as｛[ (Total - the number of items)/( the number of items×4)]×100｝with range from 0-100. A higher score indicates that the subject may be more likely to have the specific constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, Ph.D., Study Chair — China Medical University, China; Han-Kuei Wu, Ph.D., Principal Investigator — China Medical University, China; Kun San Chao, M.D., Principal Investigator — China Medical University, China; Eric Y. Chuang, Ph.D., Principal Investigator — National Taiwan University; Ming-Hsui Tsai, M.D., Principal Investigator — China Medical University, China; Yu-Chuen Huang, Ph.D., Principal Investigator — China Medical University, China; Chia-Hao Chang, M.M.S., Principal Investigator — China Medical University, China; Yao-Ching Wang, M.M.S., Principal Investigator — China Medical University, China; Chun-Hung Hua, M.D., Principal Investigator — China Medical University, China; Shih-Neng Yang, M.D., Principal Investigator — China Medical University, China; Ying-Chun Lin, M.D., Principal Investigator — China Medical University, China; Ti-Hao Wang, M.D., Principal Investigator — China Medical University, China; Ching Yun Hsieh, M.D., Principal Investigator — China Medical University, China; Ming-Yu Lien, M.D., Principal Investigator — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Hsieh HY, Yang SN, Lien MY, Wang YC, Chang CH, Wu HK, Hsu YC, Hsieh CY, Huang YC, Chang HH. Combination of Danggui Buxue Tang and concurrent chemoradiotherapy improves treatment outcomes by strengthening B cell immunity in patients with nasopharyngeal carcinoma-a double-blind, randomized trial. Transl Cancer Res. 2025 Sep 30;14(9):5199-5210. doi: 10.21037/tcr-2025-406. Epub 2025 Sep 26. PMID 41158262